CLINICAL TRIAL: NCT00512642
Title: Fluorescence Bronchoscopy and Molecular Characterization of Abnormal Bronchial Lesions: Novel Approaches for Early Detection of Lung Cancer in High Risk Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 9999999040; OH99-E-N040
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11-19

CONDITIONS: Cancer
Keywords: Cancer; Lymphocytes; Genetics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients at increased risk of lung cancer: Patients at increased risk of lung cancer

SUMMARY:
Despite intensive research efforts, there are still no simple and effective screening tools to detect early lung cancer. The majority of newly diagnosed patients have higher stage, often disseminated, non-resectable disease. A better understanding of the natural biology and molecular abnormalities in early lung lesions may aid in the development of more effective screening tools. This study will investigate the effectiveness of bronchoscopy by white light (WL) alone and in combination with Lung Imaging Fluorescence Endoscopy (LIFE) for the detection of early lung lesions in patients with a high risk for developing lung cancer. LIFE is a FDA approved adjunct to WL bronchoscopy for the screening of lung cancer and this study will provide a standardized setting in which a direct comparison between a combination of WL and LIFE versus traditional WL bronchoscopy can be made.

In addition, the study will set the stage for the collection of a unique set of biopsy specimens that will be used to learn more about the natural biology and the molecular changes in early lung lesions. We will study abnormalities in p53 by immunohistochemistry and by molecular analyses. The p53 results will be compared with histological grade and with genomic instability. Measures for genomic instability will be the loss of chromosomal information and cellular aneuploidy. Recent advances in molecular pathology, such as the development of Laser Capture Microdissection (LCM), have made the molecular profiling of these extremely small lesions feasible. The information obtained by these techniques will be used for comparison with clinical and exposure information. Future plans include the culturing of bronchial epithelial cells to study genomic instability in the multistep process of cancer progression. It is our hope that the application of these new technologies will improve the early detection of human lung cancer and provide insight into the natural biology and molecular changes of early lung lesions which may progress towards overt cancers.

DETAILED DESCRIPTION:
Despite intensive research efforts, there are still no simple and effective screening tools to detect early lung cancer. The majority of newly diagnosed patients have higher stage, often disseminated, non-resectable disease. A better understanding of the natural biology and molecular abnormalities in early lung lesions may aid in the development of more effective screening tools. The Lung Imaging Fluorescence Endoscopy (LIFE) is FDA approved as an adjunct to WL bronchoscopy for the screening of lung cancer.

Using the LIFE unit, this study will set the stage for the collection of a unique set of biopsy specimens that will be used to learn more about the natural biology and molecular changes in early lung lesions. We will study abnormalities in p53 by immunohistochemistry and by molecular analyses. The p53 results will be compared with histological grade and with genomic instability. Measures for genomic instability will be the loss of chromosomal information and cellular aneuploidy. Recent advances in molecular pathology, such as the development of Laser Capture Microdissection (LCM), have made the molecular profiling of these extremely small lesions feasible. The information obtained by these techniques will be used for comparison with clinical and exposure information. Future plans include the culturing of bronchial epithelial cells to study genomic instability in the multistep process of cancer progression. It is our hope that the application of these new technologies will improve the early detection of human lung cancer and provide insight into the natural biology and molecular changes of early lung lesions which may progress towards overt cancers.

ELIGIBILITY:
* INCLUSION CRITERIA:

Previously resected stage I, II and IIIa lung cancers.

Prior head and neck carcinoma.

Bronchogenic carcinoma in a first degree relative.

Smoking history of more than 15 pack-years current or past.

Previously treated for Hodgkin's Disease.

Abnormal sputum cytology with negative radiographs.

EXCLUSION CRITERIA:

Patients with a current clinically detectable lung cancer.

Age lower than 35 years.

Pregnant or possibly pregnant.

Patients with any contraindications to bronchoscopy.

Severe underlying medical conditions such as unstable angina, uncompensated congestive heart failure, severe airway obstruction (FEV1) less than 0.8 L), or uncontrolled hypertension.

Patients with a bleeding disorder or patients on anticoagulant therapy.

Use of chemopreventive drugs (retinoids) or photosensitizing agents (hematoporphyrin derivatives) within 3 months prior to initial bronchoscopy.

Life expectancy less than 3 months.

Patients who received chemotherapy or radiotherapy within 6 months prior to initial bronchoscopy.

Ages: 35 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 1999-07-29; Study Completion 2019-11-19

PRIMARY OUTCOMES:
Genetic abnormalities | 6 months, 12 months
  histologic or genetic change at follow-up bronchoscopy at 6 or 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jack Taylor, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] Vogelstein B, Fearon ER, Hamilton SR, Kern SE, Preisinger AC, Leppert M, Nakamura Y, White R, Smits AM, Bos JL. Genetic alterations during colorectal-tumor development. N Engl J Med. 1988 Sep 1;319(9):525-32. doi: 10.1056/NEJM198809013190901. PMID 2841597
- [Background] Lam S, MacAulay C, Hung J, LeRiche J, Profio AE, Palcic B. Detection of dysplasia and carcinoma in situ with a lung imaging fluorescence endoscope device. J Thorac Cardiovasc Surg. 1993 Jun;105(6):1035-40. PMID 8501931
- [Background] Gordenin DA, Resnick MA. Yeast ARMs (DNA at-risk motifs) can reveal sources of genome instability. Mutat Res. 1998 May 25;400(1-2):45-58. doi: 10.1016/s0027-5107(98)00047-5. PMID 9685581